CLINICAL TRIAL: NCT02829606
Title: Head Mounted Eye Tracking Aide for Loss of Central Vision
Brief Title: Head Mounted Eye Tracking Aide for Loss of Central Vision (HETALCEV)
Acronym: HETALCEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1603M84883
Record Dates: First submitted 2016-06-13; First posted 2016-07-12 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related Macular Degeneration; Central Scotoma; Head Mounted Display
MeSH Terms: conditions — Macular Degeneration; Scotoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- small scotoma using Head Mounted Display No re-mapping (Active Comparator): patients with scotoma smaller than 5 degrees NO re-mapping PLUS re-mapping
  Interventions: Other: small scotoma using Head Mounted Display No re-mapping; Other: Large scotoma using Head Mounted Display PLUS re-mapping
- Large scotoma using Head Mounted Display PLUS re-mapping (Active Comparator): patients with scotoma larger than 5 degrees NO re-mapping PLUS re-mapping
  Interventions: Other: small scotoma using Head Mounted Display No re-mapping; Other: Large scotoma using Head Mounted Display PLUS re-mapping

INTERVENTIONS:
Other: small scotoma using Head Mounted Display No re-mapping — re-mapping software turned off
Other: Large scotoma using Head Mounted Display PLUS re-mapping — re-mapping software turned on

SUMMARY:
A device has been developed that has eye trackers integrated within the Head Mounted Display (HMD) and can remap text and images around the scotoma in real time to prevent information loss from a central scotoma. It can also carry out other types of image processing such as contrast enhancement and image magnification. The aim of this study is to assess the efficacy of this device on the visual performance of participants suffering from central vision loss, with and without remapping

DETAILED DESCRIPTION:
Participants with bilateral central scotomas will be selected for this study during their routine clinical visits at the University of Minnesota Eye Clinic. Written consent will be obtained from all participants.

Each participant will have their scotomas mapped using a Nidek MP-1 microperimeter housed in the psychology department to give exact size and shape information. This allows for the extent of each eye's scotoma to be put into the remapping software, and their intersection used in remapping calculation. Comparisons will be made between participants with small scotoma, less than 5 degrees, and participants with large scotoma, larger than 5 degrees. Experiments to be performed with the device are also divided into two categories. Category 1 involves reading of naturalistic text, and everyday task performance. Category 2 involves studying the effects of practice with the device on performance in category 1 experiments.

Participants will schedule an initial one-hour session for testing. During testing, participants will be told about the device and its functionality. Main instructions include what patients can expect to experience and see when wearing the HMD. Following this, the participants will be instructed on how to wear the HMD. If they have any glasses/ corrective lenses, they can be kept on. Once the patients don the HMD, testing will begin.

Initially, a calibration-free mode will be tested. This will entail asking the subject to focus on a particular point on the screen and checking if the gaze point determined by the eye tracker corresponds to this point. If good calibration is obtained, the investigators proceed with testing. Otherwise, a 3-point calibration sequence will be initiated following instructions on the software program. For the 3-point calibration sequence, the participant will be instructed to fixate at 3-5 different points on the screen one at a time. Following this calibration sequence, testing will resume and visual performance such as reading speed in words/minute will be measured as the primary outcome measure, with and without remapping.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Central vision loss from bilateral central scotomas
* No cognitive impairment as indicated by a Mini-Mental State Examination (MMSE)

Exclusion Criteria:

* Failed MMSE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Reading speed | 5 years
  words/minute

CONTACTS AND LOCATIONS:
Overall Officials: Erik van Kuijk, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University _of_Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
participants will be de-identified